CLINICAL TRIAL: NCT01666587
Title: The Role of Prostaglandin and Anti-oxidant Availability on Recovery From Forearm Ischemia-reperfusion Injury in Humans
Brief Title: Ischemia Reperfusion: Prostaglandins and Antioxidants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Essex (Other)
Responsible Party: Principal Investigator, Mark Rakobowchuk, Principle Investigator, University of Essex
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRAPC; DBD0300 (Other: Biological Sciences)
Record Dates: First submitted 2012-08-09; First posted 2012-08-16 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Ischemic Reperfusion Injury
MeSH Terms: interventions — Antioxidants; Prostaglandin Antagonists; Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control (No Intervention): Control trial to determine the impact of the ischemic injury on vascular function without intervention
- Antioxidant load (Experimental): Trial to determine the impact of an antioxidant load before the ischemic injury on vascular function recovery
  Interventions: Dietary Supplement: Antioxidant
- Prostaglandin inhibition (Experimental): Trial to determine the impact of a non-selective prostaglandin inhibitor before the ischemic injury on vascular function recovery
  Interventions: Drug: Prostaglandin inhibitor (Ibuprophen)
- Combined (Experimental): Trial to determine the impact of an antioxidant load and prostaglandin inhibitor before the ischemic injury on vascular function recovery
  Interventions: Dietary Supplement: Antioxidant; Drug: Prostaglandin inhibitor (Ibuprophen)

INTERVENTIONS:
Dietary Supplement: Antioxidant
  Arms: Antioxidant load; Combined
Drug: Prostaglandin inhibitor (Ibuprophen)
  Other Names: ibuprofen
  Arms: Combined; Prostaglandin inhibition

SUMMARY:
The purposes of this study are two-fold. The first purpose is to determine the effect of taking vitamins on the recovery of an artery (blood vessel) following an induced temporary injury. The second purpose is to determine whether a specific vasodilator is less abundant after the injury and whether this contributes to increased constriction or after the injury. Finally, does vitamin consumption have an effect on the recovery from the injury if one of the substances in the blood that causes vessels to enlarge (dilate) is stopped?

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Healthy females

Exclusion Criteria:

* Smokers
* Cardiovascular disease
* Peripheral vascular disease
* Neurological deficits
* Diabetes Type I or II
* Pregnant women
* Adverse reactions to Ibuprofen

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in flow mediated dilation | Change from baseline at 15 minutes after ischemia-reperfusion injury
  Flow mediated dilation is a measure of vascular function and is measured as the outcome before and after an injury to the inner lining of the artery.

SECONDARY OUTCOMES:
Change in low flow mediated constriction | Change from baseline at 15 minutes after ischemia-reperfusion injury
  low flow mediated constriction is a measure of vascular function and is measured to establish the impact of a vascular injury

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rakobowchuk, PhD, Principal Investigator — Thompson Rivers University
Locations (1):
- University of Essex, Colchester, Essex, United Kingdom